CLINICAL TRIAL: NCT01475851
Title: A Multi-center, Open-label Study of GSK548470 (Tenofovir Disoproxil Fumarate) in Patients With Compensated Chronic Hepatitis B With Poor Response to Other Drugs
Brief Title: Phase 3 Study of GSK548470 in Patients With Compensated Chronic Hepatitis B With Poor Response to Other Drugs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115912
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Results first posted 2013-11-04 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-05

CONDITIONS: Hepatitis B, Chronic
Keywords: Tenofovir disoproxil fumarate, compensated chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK548470 300 mg (Experimental): GSK548470 300 mg tablet is administered orally once daily
  Interventions: Drug: GSK548470 300 mg tablet

INTERVENTIONS:
Drug: GSK548470 300 mg tablet — Blue tablets containing 300 mg of tenofovir disoproxil fumarate
  Other Names: GSK548470

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of once-daily treatment with GSK548470 300 mg in Japanese patients with compensated chronic hepatitis B with poor response to other drugs.

DETAILED DESCRIPTION:
This is a multicenter, open-label study in Japanese patients with compensated chronic hepatitis B with poor response to other drugs in order to evaluate the efficacy and safety of GSK548470 administered at a dose of 300 mg once daily. The target sample size is set at 32 subjects. The primary objective is to evaluate the efficacy and safety of once-daily treatment with GSK548470 300 mg in subjects with compensated chronic hepatitis B with poor response to other drugs. The secondary objective is to evaluate the long-term efficacy and safety of once-daily treatment with GSK548470 300 mg.To evaluate the efficacy and safety of GSK548470 in the study, subjects receiving a combination of lamivudine (LAM) and adefovir pivoxil (ADV) will be switched to a combination of LAM and GSK548470, while subjects on entecavir hydrate (ETV) with or without ADV will be switched to a combination of ETV and GSK548470.

ELIGIBILITY:
Inclusion Criteria:

* The ability to understand and sign a written informed consent form
* 16 to 69 years of age at the time of informed consent
* Females of childbearing potential must have a negative pregnancy test and agree to avoidance of pregnancy
* Subject must show QTc <450 millisecond (msec) or <480msec with Bundle Branch Block
* Chronic HBV infection, defined as positive serum HBsAg for at least 6 month
* Subjects currently treated with LAM/ADV, ETV or ETV/ADV for greater than 24 weeks
* Chronic hepatitis B ; HBV NDA >= 4 log10 copies/mL, Chronic hepatitis B with cirrhosis ; HBV NDA >= 3 log10 copies/mL
* Serum ALT <= 10 × ULN
* Creatinine clearance >= 70 mL/min
* Haemoglobin >= 8 g/dL
* WBC >= 1,000 /mm3

Exclusion Criteria:

* Decompensated liver disease
* Co-infection with HIV or HCV
* Autoimmune hepatitis rather than chronic hepatitis B
* Subject with serious complication
* Received or have a plan for solid organ or bone marrow transplantation
* Has proximal tubulopathy
* History of hypersensitivity to nucleoside and/or nucleotide analogues
* Evidence of hepatocellular carcinoma by diagnostic imaging at screening and/or serum α-fetoprotein > 50 ng/mL at screening
* History of HCC
* Received any interferon or HB vaccine therapy within 24 weeks prior to initiation
* Received overdose NSAIDs, excluding temporary or topical use, within 7 days prior to initiation
* Received drugs for injection containing glycyrrhizin as the main component within 4 weeks prior to initiation
* Received drugs causing renal impairment, competitors of renal excretion, immunosuppressants, chemotherapeutics and/or corticosteroids within 8 weeks prior to initiation
* Participation in another clinical study within 6 months of study entry or planned participation in another clinical study after entry to this study
* Woman who is pregnant, lactating, possibly pregnant or planning a pregnancy during the study period
* Psychiatry disorder or cognitive disorder that may affect the subject ability to give informed consent or to follow specified study procedures
* History of alcohol or drug abuse
* Any condition or situation that may interfere with the subject's participation in the study

Ages: 16 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Japan (9):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Tokyo

REFERENCES:
- [Derived] Kumada H, Koike K, Suyama K, Ito H, Itoh H, Sugiura W. Efficacy and safety of tenofovir disoproxil fumarate rescue therapy for chronic hepatitis B patients who failed other nucleos(t)ide analogs. Hepatol Res. 2017 Sep;47(10):1032-1041. doi: 10.1111/hepr.12842. Epub 2016 Dec 21. PMID 27862721

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 34 participants (13 participants in the Lamivudine [LAM]/ Tenofovir disoproxil fumarate [TDF] group and 21 participants in the Entecavir [ETV]/TDF group) were enrolled in the study
Groups:
- LAM 100 mg/TDF 300 mg: Participants received a single, Open-Label (OL) Lamivudine (LAM) 100 milligram (mg) tablet once daily (OD) and a single, OL tenofovir disoproxil fumarate (TDF) 300 mg tablet OD for 96 weeks.
- ETV 0.5 mg/TDF 300 mg: Participants received a single, OL entecavir (ETV) 0.5 mg tablet OD and a single, OL TDF 300 mg tablet OD for 96 weeks.
Period: Overall Study
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg
Started | 13 | 21
Completed | 12 | 21
Not Completed | 1 | 0
Not completed — Protocol defined stopping criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg | Total
Number analyzed (Participants) | 13 | 21 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.1 (7.57) | 50.3 (9.18) | 51.0 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 17 | 25
Race/Ethnicity, Customized [Number; unit: Participants] — HER=Heritage
  Participants
    Asian-Japanese Heritage | 13 | 21 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HBV DNA Level < 2.1 log10 Copies/mL at Week 24
Description: The number of participants with serum hepatitis B virus deoxyribonucleic acid (HBV DNA) level < the lower limit of quantitation (2.1 log10 copies/millilitres[copies/mL]) (i.e., the rate of suppression) at Week 24 was summarized. Statistical analysis was not provided for the number of participants achieving HBV DNA <2.1 log10 copies/mL (at Week 24). Missing values observed during the treatment period was imputed by the last observation carried forward (LOCF) method.
Time Frame: Week 24
Population: Full Analysis Set (FAS) Population: all participants who received at least one dose of investigational product (IP) and had at least one efficacy assessment after the start of study treatment.
Measure: Number; unit: participants
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg
Number analyzed (Participants) | 13 | 21
participants | 8 | 12

2. Secondary Outcome: Mean Change From Baseline in Serum HBV DNA Level at Week 24, Week 48 and Week 96
Description: The mean change from Baseline in the hepatitis B virus deoxyribonucleic acid (HBV DNA) level at Week 24, Week 48 and Week 96 were assessed (HBV DNA values below the lower limit of quantitation [i.e. 2.1 log10 copies/mL] for the assay were set to the lower limit minus 0.1 [i.e. 2.0 log10 copies/mL]). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Last Observation Carried Forward (LOCF) method was applied for missing values.
Time Frame: Baseline and Week 24, Week 48 and Week 96
Population: FAS Population
Measure: Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg
Number analyzed (Participants) | 13 | 21
log10 copies/mL
  Week 24 | -2.72 [-3.50 to -1.93] | -3.33 [-4.01 to -2.65]
  Week 48 | -2.88 [-3.70 to -2.06] | -3.50 [-4.28 to -2.73]
  Week 96 | -3.02 [-3.84 to -2.21] | -3.50 [-4.35 to -2.66]

3. Secondary Outcome: Number of Participants With Serum HBV DNA < 2.1 log10 Copies/mL at Week 48 and Week 96
Description: The number of participants with serum HBV DNA level < the lower limit of quantitation (2.1 log10 copies/mL) (i.e., the rate of suppression) at Week 48 and Week 96 were summarized. The LOCF method was applied for missing values.
Time Frame: Week 48 and Week 96
Population: FAS Population.
Measure: Number; unit: participants
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg
Number analyzed (Participants) | 13 | 21
participants
  Week 48 | 9 | 12
  Week 96 | 10 | 14

4. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) Normalization at Week 24, Week 48 and Week 96
Description: The number of participants with alanine aminotransferase (ALT) normalization at Week 24, Week 48 and Week 96 were summarized. ALT normalization is defined as when an ALT value exceeds the upper limit of normal range (ULN) at Baseline and within the normal range at the end of treatment. The LOCF method was applied for missing values.
Time Frame: Week 24, Week 48 and Week 96
Population: Biochemically Evaluable Population (BEP): all participants who received at least one dose of investigational product and with an abnormal ALT at Baseline. The population for the analysis of ALT normalization was all participants with an ALT value > ULN at Baseline.
Measure: Number; unit: participants
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg
Number analyzed (Participants) | 5 | 10
participants
  Week 24 | 3 | 6
  Week 48 | 3 | 5
  Week 96 | 3 | 6

5. Secondary Outcome: Number of Participants With HBeAg Loss at Week 24, Week 48 and Week 96
Description: The number of participants achieving hepatitis Be antigen (HBeAg) loss at Week 24, Week 48 and Week 96 in positive HBeAg participants at Baseline were summarized. Loss of HBeAg is defined as the change of detectable HBeAg from positive to negative. The LOCF method was applied for missing values.
Time Frame: Week 24, Week 48 and Week 96
Population: FAS Population
Measure: Number; unit: participants
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg
Number analyzed (Participants) | 11 | 17
participants
  Week 24 | 0 | 0
  Week 48 | 1 | 0
  Week 96 | 1 | 0

6. Secondary Outcome: Number of Participants With HBeAg/HBeAb Seroconversion at Week 24, Week 48 and Week 96
Description: The number of participants achieving hepatitis Be antigen (HBeAg)/hepatitis B e antibody (HBeAb) seroconversion at Week 24, Week 48 and Week 96 in positive HBeAg and negative HBeAb participants at Baseline were summarized. Seroconversion to HBeAg is defined as change of detectable antibody to HBeAg from negative to positive. The LOCF method was applied for missing values.
Time Frame: Week 24, Week 48 and Week 96
Population: FAS Population
Measure: Number; unit: participants
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg
Number analyzed (Participants) | 11 | 17
participants
  Week 24 | 0 | 0
  Week 48 | 0 | 0
  Week 96 | 0 | 0

7. Secondary Outcome: Number of Participants Achieving HBsAg Loss at Week 24, Week 48 and Week 96
Description: The number of participants with hepatitis B surface antigen (HBsAg) loss at Week 24, Week 48 and Week 96 in positive HBsAg participants at Baseline were summarized. Loss of HBsAg is defined as change of detectable HBsAg from positive to negative. The LOCF method was applied for missing values.
Time Frame: Week 24, Week 48 and Week 96
Population: FAS Population
Measure: Number; unit: participants
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg
Number analyzed (Participants) | 13 | 21
participants
  Week 24 | 0 | 0
  Week 48 | 0 | 0
  Week 96 | 0 | 0

8. Secondary Outcome: Number of Participants Achieving HBsAg/HBsAb Seroconversion at Week 24, Week 48 and Week 96
Description: The number of participants with hepatitis B surface antigen (HBsAg)/hepatitis B surface antibody (HBsAb) seroconversion at Week 24, Week 48 and Week 96 in positive HBsAg and negative HBsAb participants at Baseline were summarized. HBsAg seroconversion was defined as change of detectable antibody to HBsAg from negative to positive. The LOCF method was applied for missing values.
Time Frame: Week 24, Week 48 and Week 96
Population: FAS Population
Measure: Number; unit: participants
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg
Number analyzed (Participants) | 13 | 21
participants
  Week 24 | 0 | 0
  Week 48 | 0 | 0
  Week 96 | 0 | 0

9. Secondary Outcome: Number of Participants With Virological Breakthrough and Resistance-related Mutations
Description: The number of participants who harbored resistance-related mutations and developed virological breakthrough was summarized. Virological breakthrough defined as HBV DNA level increase >=1 log10 copies/mL above the treatment nadir were analyzed through end of treatment. Subjects who achieved the HBV-DNA values below lower limit of quantification (LLQ) (< 2.1 log10 copies/mL) in quantitative analysis at Week 96 were also considered "negative" in drug-resistance without implementation of genotypic analysis. Lamivudine (LAM), adefovir pivoxil (ADV), and entecavir hydrate (ETV) resistance-related mutations were analyzed at Screening (i.e. Baseline), Week 24, Week 48 and Week 96 in participants with HBV DNA level above the lower limit of detection. Virologic breakthrough was defined as 1.0 log10 or greater increases in serum HBV DNA levels from on-treatment nadir. The LOCF method was applied for missing values.
Time Frame: Screening, Week 24, Week 48, Week 96 and Virological Breakthrough
Population: FAS Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Number; unit: participants
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg
Number analyzed (Participants) | 13 | 21
participants
  Virological breakthrough, through end of study n=0 | 0 | 1
  LAM resistance-related mutations,Screening,n=13,21 | 11 | 17
  ADV resistance-related mutations,Screening,n=13,21 | 4 | 0
  ETV resistance-related mutations,Screening,n=13,21 | 6 | 16
  LAM resistance-related mutations, Week 24, n=5, 9 | 4 | 8
  ADV resistance-related mutations, Week 24, n=5, 9 | 2 | 0
  ETV resistance-related mutations, Week 24, n=5, 9 | 1 | 8
  LAM resistance-related mutations, Week 48, n= 3, 9 | 2 | 7
  ADV resistance-related mutations, Week 48, n= 3, 9 | 1 | 0
  ETV resistance-related mutations, Week 48, n= 3, 9 | 1 | 7
  LAM resistance-related mutations, Week 96, n= 2, 7 | 2 | 6
  ADV resistance-related mutations, Week 96, n= 2, 7 | 1 | 0
  ETV resistance-related mutations, Week 96, n= 2, 7 | 2 | 6
  LAM resistance-related mutations, VB, n=0,1 | 0 | 1
  ADV resistance-related mutations, VB, n=0,1 | 0 | 0
  ETV resistance-related mutations, VB, n=0,1 | 0 | 1

10. Secondary Outcome: Number of Participants Achieving Each Indicated HBsAg Category at Baseline, Week 24, Week 48 and Week 96
Description: The number of participants achieving each indicated hepatitis B surface antigen (HBsAg) category (HBsAg <80, 80 to 800, 800 to 8000, 8000 to 80000, >=80000) (kilo international unit per liter [KIU/L]) by study visit was summarized.
Time Frame: Baseline, Week 24, Week 48 and Week 96
Population: FAS Population
Measure: Number; unit: participants
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg
Number analyzed (Participants) | 13 | 21
participants
  HBsAg <80 KIU/L, Baseline | 0 | 0
  HBsAg 80-800 KIU/L, Baseline | 1 | 0
  HBsAg 800-8000 KIU/L, Baseline | 6 | 12
  HBsAg 8000-80,000 KIU/L, Baseline | 6 | 8
  HBsAg >=80,000 KIU/L, Baseline | 0 | 1
  HBsAg <80 KIU/L, Week 24 | 0 | 0
  HBsAg 80-800 KIU/L, Week 24 | 3 | 0
  HBsAg 800-8000 KIU/L, Week 24 | 5 | 15
  HBsAg 8000-80,000 KIU/L, Week 24 | 5 | 6
  HBsAg >=80,000 KIU/L, Week 24 | 0 | 0
  HBsAg <80 KIU/L, Week 48 | 0 | 0
  HBsAg 80-800 KIU/L, Week 48 | 3 | 1
  HBsAg 800-8000 KIU/L, Week 48 | 5 | 14
  HBsAg 8000-80,000 KIU/L, Week 48 | 5 | 6
  HBsAg >=80,000 KIU/L, Week 48 | 0 | 0
  HBsAg <80 KIU/L, Week 96 | 0 | 0
  HBsAg 80-800 KIU/L, Week 96 | 4 | 3
  HBsAg 800-8000 KIU/L, Week 96 | 6 | 13
  HBsAg 8000-80,000 KIU/L, Week 96 | 3 | 5
  HBsAg >=80,000 KIU/L, Week 96 | 0 | 0

11. Secondary Outcome: Number of Participants Achieving Each Indicated HBcrAg Category at Baseline,Week 24, Week 48 and Week 96
Description: The number of participants achieving each indicated hepatitis B core-related antigen (HBcrAg) category (HBcrAg <3.0 log10, 3.0 to 4.0 log10, 4.0 to 5.0 log10, 5.0 to 6.0 log10, >=6.0 log10) (kilo units per liter [KU/L]) by study visit was summarized. The LOCF method was applied for missing values.
Time Frame: Baseline, Week 24, Week 48 and Week 96
Population: FAS Population
Measure: Number; unit: Participants
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg
Number analyzed (Participants) | 13 | 21
Participants
  HBcrAg <3.0 Log KU/L, Baseline | 0 | 0
  HBcrAg 3.0-4.0 Log KU/L, Baseline | 0 | 1
  HBcrAg 4.0-5.0 Log KU/L, Baseline | 0 | 1
  HBcrAg 5.0-6.0 Log KU/L, Baseline | 1 | 0
  HBcrAg >=6.0 Log KU/L, Baseline | 12 | 19
  HBcrAg <3.0 Log KU/L, Week 24 | 0 | 0
  HBcrAg 3.0-4.0 Log KU/L, Week 24 | 0 | 1
  HBcrAg 4.0-5.0 Log KU/L, Week 24 | 1 | 1
  HBcrAg 5.0-6.0 Log KU/L, Week 24 | 1 | 1
  HBcrAg >=6.0 Log KU/L, Week 24 | 11 | 18
  HBcrAg <3.0 Log KU/L, Week 48 | 0 | 0
  HBcrAg 3.0-4.0 Log KU/L, Week 48 | 1 | 1
  HBcrAg 4.0-5.0 Log KU/L, Week 48 | 0 | 1
  HBcrAg 5.0-6.0 Log KU/L, Week 48 | 2 | 1
  HBcrAg >=6.0 Log KU/L, Week 48 | 10 | 18
  HBcrAg <3.0 Log KU/L, Week 96 | 0 | 0
  HBcrAg 3.0-4.0 Log KU/L, Week 96 | 1 | 1
  HBcrAg 4.0-5.0 Log KU/L, Week 96 | 0 | 1
  HBcrAg 5.0-6.0 Log KU/L, Week 96 | 3 | 2
  HBcrAg >=6.0 Log KU/L, Week 96 | 9 | 17

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication to the end of the treatment period (up to average of 96 weeks).
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who received at least one dose of investigational product.
Arm/Group | LAM 100 mg/TDF 300 mg | ETV 0.5 mg/TDF 300 mg
Serious Adverse Events (participants affected / at risk) | 1/13 | 2/21
Other Adverse Events (participants affected / at risk) | 12/13 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAM 100 mg/TDF 300 mg (N=13) | ETV 0.5 mg/TDF 300 mg (N=21)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LAM 100 mg/TDF 300 mg (N=13) | ETV 0.5 mg/TDF 300 mg (N=21)
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Dysaesthesia (Nervous system disorders) | 1 | 2
Parosmia (Nervous system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 7 | 11
Otitis externa (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3
Asparatate aminotransferase increased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2
Fatigue (General disorders) | 0 | 2
Malaise (General disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 3
Gallbladder polyp (Hepatobiliary disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.